CLINICAL TRIAL: NCT04493983
Title: Evaluation of Oxidative Stress-related Biomarkers With a Histopathological and Biochemical Approach in Ovarian Tissue From a Human Carbondioxide Pneumoperitoneum-applied Ischemia/Reperfusion Model
Brief Title: Role of Oxidative Stress in Ovarian Tissue After CO2-pneumoperitoneum Application-induced I/R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ismet Hortu (Other)
Responsible Party: Sponsor-Investigator, Ismet Hortu, Clinical researcher, Ismet Hortu, MD., PhD. Department of Obstetrics and Gynecology, Ege University School of Medicine, Izmir, Turkey, Ege University
Organization: Ege University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7-11/62
Record Dates: First submitted 2020-07-26; First posted 2020-07-30 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Oophorectomy; Oxidative Stress; Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigation (Other): Unilateral oophorectomy was performed immediately after abdominal entry, and the remaining contralateral ovary was excised at the end of the hysterectomy in order to compare the effect of these surgical procedures on ovarian tissue.
  Interventions: Procedure: laparoscopic salpingo-oophorectomy; Procedure: Laparoscopic bilateral salpingo-oophorectomy

INTERVENTIONS:
Procedure: laparoscopic salpingo-oophorectomy — Laparoscopic bilateral salpingo-oophorectomy
Procedure: Laparoscopic bilateral salpingo-oophorectomy — Unilateral oophorectomy was performed immediately after abdominal entry, and the remaining contralateral ovary was excised at the end of the hysterectomy in order to compare the effect of these surgical procedures on ovarian tissue.

SUMMARY:
Because of cellular changes in response to ischemia and a following period of reperfusion, damages to organs and different tissues occur. There are several ongoing studies to enlighten the pathophysiological processes underlying these damages inflicted by ischemia/reperfusion.

Gases (CO2) with low water content are used in pneumoperitoneum, which is a procedure to inflate the abdominal cavity with an appropriate gas for laparoscopic operations. In the current literature, it was shown that due to a restricted blood flow during the gas insufflation, ischemia develops and with the reperfusion of the organ in deflation period, oxidative stress and inflammation increases, leading to ischemia/reperfusion-related organ and tissue damages.

In the proposed study, biomarkers for ischemia/reperfusion-inflicted damage will be evaluated in a biochemical and histopathological perspective in biopsy samples of ovaries from a young patient group in which hysterectomy and bilateral salpingo-oophorectomy will be performed, laparoscopically.

DETAILED DESCRIPTION:
In the laparoscopic salpingo-oophorectomy, after the induction of anesthesia, an umbilical skin incision was performed. Pneumoperitoneum was established using dry, nonheated CO2 insufflation through a Veress needle. A 10-mm trocar was inserted into the abdominal cavity through the umbilical incision for the laparoscope. Subsequently, three 5-mm ancillary trocars, 2 on the lower abdominal quadrants and 1 on the left upper quadrant, were introduced to the abdominal space under direct optic visualization. IAP was set at 14 mm Hg and maintained with a gas insufflator (Endoflator; Karl Storz Endoscopy, Tuttlingen, Germany)Immediately after the port placement, unilateral oophorectomy was performed, and ovarian biopsies were obtained. The operation continued with ligation and transection of the contralateral utero-ovarian ligament and the bilateral round ligaments. The contralateral infundibulopelvic ligament, which contains the main vascular supply for the contralateral ovary, remained intact. Subsequently, anterior and posterior leaflets of the broad ligament were identified and dissected, and the bladder was placed away from the lower uterine segment. The uterus removed from vaginal way after necessary steps. After desufflation, the cuff closure procedure was performed vaginally. At the end of the closure, pneumoperitoneum was reestablished, the remaining contralateral ovary was removed immediately, and biopsies were obtained for histologic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Transgender Men who wants to remove their uterus and both ovaries.

Exclusion Criteria:

* Known endometriosis
* Hysterectomized patient
* Unacceptance to involve to the trial
* Suspicion of malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Impact of CO2 pneumoperitoneum on ovaries by comparing histopathology | 1-day (at the time of the surgery)
  Histopathological investigation of ovaries after CO2 pneumoperitoneum -induced I/R

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University School of Medicine, Department of Obstetrics and Gynecology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guven S, Muci E, Unsal MA, Yulug E, Alver A, Kadioglu Duman M, Mentese A. The effects of carbon dioxide pneumoperitoneum on ovarian blood flow, oxidative stress markers, and morphology during laparoscopy: a rabbit model. Fertil Steril. 2010 Mar 1;93(4):1327-32. doi: 10.1016/j.fertnstert.2008.10.053. Epub 2008 Dec 9. PMID 19081089
- [Result] Schafer M, Krahenbuhl L. Effect of laparoscopy on intra-abdominal blood flow. Surgery. 2001 Apr;129(4):385-9. doi: 10.1067/msy.2001.110224. No abstract available. PMID 11283527
- [Result] Cevrioglu AS, Yilmaz S, Koken T, Tokyol C, Yilmazer M, Fenkci IV. Comparison of the effects of low intra-abdominal pressure and ischaemic preconditioning on the generation of oxidative stress markers and inflammatory cytokines during laparoscopy in rats. Hum Reprod. 2004 Sep;19(9):2144-51. doi: 10.1093/humrep/deh380. Epub 2004 Jun 30. PMID 15229201
- [Result] Biler A, Yucebilgin S, Sendag F, Akman L, Akdemir A, Ates U, Uyanikgil Y, Yilmaz-Dilsiz O, Sezer E. The effects of different intraabdominal pressure protocols in laparoscopic procedures on oxidative stress markers and morphology in rat ovaries. Adv Clin Exp Med. 2014 Nov-Dec;23(6):885-92. doi: 10.17219/acem/37331. PMID 25618113
- [Result] Akdemir A, Taylan E, Sahin C, Ozgurel B, Karlitepe A, Zekioglu O, Ercan G. The Impact of Carbon Dioxide Pneumoperitoneum on Ovarian Ischemia-Reperfusion Injury during Laparoscopic Surgery: A Preliminary Study. J Minim Invasive Gynecol. 2018 May-Jun;25(4):638-643. doi: 10.1016/j.jmig.2017.10.018. Epub 2017 Nov 28. PMID 29107119